CLINICAL TRIAL: NCT03362541
Title: A Multi-Site Randomized Controlled Trial of MS INFoRm: An Interactive Fatigue Management Resource for Persons With Multiple Sclerosis
Brief Title: A Multi-Site Trial of MS INFoRm (Fatigue Management Resource)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Marcia Finlayson (Other)
Collaborators: University of Alberta (Other); University of Calgary (Other)
Responsible Party: Sponsor-Investigator, Dr. Marcia Finlayson, Vice Dean Health Sciences, Director School of Rehabilitation Therapy, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6020674
Record Dates: First submitted 2017-11-20; First posted 2017-12-05 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; fatigue; self-management; rehabilitation
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Intervention Model Description: This study will use a randomized controlled trial design to test the efficacy and effectiveness of MS INFoRm. Two hundred participants from at least three sites across Canada will be randomly assigned to one of two groups: the experimental (MS INFoRm) group or usual care control group. After completing the study, participants in the usual care control group will be given access to MS INFoRm in order to provide them with any benefits of the website, if any are uncovered. Both groups will be evaluated on primary (fatigue impact) and secondary (self-efficacy, cognitive function, participation and autonomy, depression) outcomes at baseline (week 1), after 3-month use of the MS INFoRm website (week 12), and after 6-month follow-up (week 36).
Who Masked: Participant, Outcomes Assessor
Masking Description: Both the MS INFoRm group and the control group will receive a login and password, although participants in the groups will be directed to a different webpages (i.e. a MS INFoRm page or usual care control webpage). This will facilitate blinding of participants to their allocation. The research assistant will complete the scheduling, data collection, and data entry blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MS INFoRm group (Experimental): Participants in the MS INFoRm group will be given a login and password that will take them to the MS INFoRm webpage. Access will be granted for 3-months, starting on the date of the first login. Participants can access the website at any time, at their own volition over the 3-months.
  Interventions: Behavioral: MS INFoRm
- Usual care control group (Active Comparator): Participants in the usual care group will be given a login and password that will take them to a usual care webpage. Access will be granted for 3-months, starting on the date of the first login. Participants can access the website at any time, at their own volition over the 3-months.
  Interventions: Behavioral: Usual Care Control Group

INTERVENTIONS:
Behavioral: MS INFoRm — MS INFoRm incorporates principles of self-management and adult learning theory. The contents address the sources of fatigue, ways of monitoring fatigue, and strategies to reduce fatigue.
  Arms: MS INFoRm group
Behavioral: Usual Care Control Group — The usual care webpage will contain content from widely available resources about MS fatigue.
  Arms: Usual care control group

SUMMARY:
People with MS commonly experience extreme fatigue that negatively impacts their ability to engage in a full range of daily activities, quality of life, and employment. A new website called MS INFoRm (Multiple Sclerosis: An Interactive Fatigue Management Resource) allows people with MS to take a personalized and active approach to learning about and managing their fatigue. The aims of this study are:

1. To determine to determine whether 3-month use of the MS INFoRm website can reduce the impact of fatigue on daily life among persons with MS.
2. To determine whether 3-month use of the MS INFoRm website results in improvement in self- efficacy/ confidence for managing MS fatigue, self-reported cognitive function, participation and autonomy/ independence, and depression.
3. To determine whether benefits are maintained among the MS INFoRm users after 6-months.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of MS
* between 18 and 65 years of age
* access to a computer or other electronic device with internet access on which to use the website
* report mild to moderate fatigue
* live in Canada

Exclusion Criteria:

* any major comorbid conditions that might influence fatigue management (lupus, rheumatoid arthritis, chronic obstructive lung disease, chronic fatigue syndrome)
* report difficulty reading and comprehending English written at a Grade 7 level
* report upper extremity or visual impairments that cannot be accommodated adequately to enable computer access

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Change in the Modified Fatigue Impact Scale | Administered at baseline (week 1), 3-months (week 12), and 6-months (week 36).
  21-item scale which assesses the impact of fatigue on daily functioning during the last four weeks.

SECONDARY OUTCOMES:
Change in the Multiple Sclerosis Self-Efficacy Scale | Administered at baseline (week 1), 3-months (week 12), and 6-months (week 36).
  14-item scale measuring self-efficacy in which respondents rate the degree to which they believe they can overcome challenges.
Change in the Perceived Deficits Questionnaire | Administered at baseline (week 1), 3-months (week 12), and 6-months (week 36).
  20-item questionnaire assessing perceived cognitive function across the domains most commonly affected in MS: attention, retrospective memory, prospective memory, and planning and organization.
Change in the Center for Epidemiological Studies Depression Scale | Administered at baseline (week 1), 3-months (week 12), and 6-months (week 36).
  20-item scale which assesses depressive symptomatology.
Change in the Impact on Participation and Autonomy Questionnaire | Administered at baseline (week 1), 3-months (week 12), and 6-months (week 36).
  Provides a measure of limitations in participation and autonomy. The tool includes 39 questions across 5 domains: autonomy indoors, autonomy outdoors, family role, social life and relationships, and work and education.

CONTACTS AND LOCATIONS:
Overall Officials: Marcia Finlayson, PhD, Principal Investigator — Queen's University
Locations (3):
- Canada (3):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Queen's University, Kingston, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Finlayson M, Akbar N, Turpin K, Smyth P. A multi-site, randomized controlled trial of MS INFoRm, a fatigue self-management website for persons with multiple sclerosis: rationale and study protocol. BMC Neurol. 2019 Jun 25;19(1):142. doi: 10.1186/s12883-019-1367-6. PMID 31238966